CLINICAL TRIAL: NCT06254846
Title: Evaluation of First-void Urine as an Alternative to Cervical Sampling for Human Papillomavirus (HPV) Testing in Cervical Cancer Screening (Single-center Study).
Acronym: URAPREV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23CH137; 2023-A02247-38 (Other: ANSM)
Record Dates: First submitted 2024-01-29; First posted 2024-02-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Uterine Cervical Cancer
Keywords: HPV; Cervical cancer; Cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre study to assess the diagnostic performance (sensitivity and specificity) of HPV PCR on 1st-draft urine compared with cervico-vaginal sampling (= gold standard).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary screening for UCC (Other): Women aged between 30 and 65 who are candidates for primary screening for UCC will be included.
  Interventions: Other: Urine sample, 1st stream; Other: Cervico-vaginal swab

INTERVENTIONS:
Other: Urine sample, 1st stream — Use of the Colli-Pee® device for collecting the first urine stream
Other: Cervico-vaginal swab — Use of a "gold standard" reference method = HPV PCR using the Anyplex® II HPV HR kit (Seegene) carried out on a cervico-vaginal swab in ThinPrep® medium (liquid medium medium into which the cervico-vaginal swab is discharged).

SUMMARY:
Papillomaviruses are responsible for almost all cervical cancers. In France, there are more than 3000 new cases of cervical cancer each year and nearly 1000 deaths. One of the ways to prevent this cancer is screening by PCR on cervical sample for which national coverage rate remains very insufficient (<60%). The invasive and uncomfortable nature of cervical sampling has been identified as a major obstacle to screening. In this context, an alternative sample, such as the first-void urine, seems to be judicious. Nevertheless, some studies have shown a lack of sensitivity of the HPV PCR test on urine. As underlined by the French National Authority for Health (HAS), this is mainly due to a lack of standardization of urine collection. In this study, the investigators therefore propose to evaluate the performance of the HPV PCR test on first-void urine using a standardized protocol. Through a questionnaire, they will also evaluate the acceptability of the first void urine collection device.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age between 30 and 65
* Consulting in the Gynecology-Obstetrics department for primary cervical cancer screening
* Patient affiliated or entitled to a social security regimen
* Patient who has received information about the study and expressed non-opposition

Exclusion Criteria:

-

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
specificity | Month : 12
  specificity (%) of the HPV PCR test on the first void urine (Colli-Pee®) in comparison with the same HPV PCR test applied to the cervical sampling (= gold standard).
Sensitivity | Month : 12
  Sensitivity (%) of the HPV PCR test on the first void urine (Colli-Pee®) in comparison with the same HPV PCR test applied to the cervical sampling (= gold standard).

SECONDARY OUTCOMES:
HPV genotype concordance | Month : 12
  Percentage of HPV genotype concordance between first void urine and cervical sample.
Women with a positive evaluation | Month : 12
  Percentage of women with a positive evaluation of the first void urine collection device.

CONTACTS AND LOCATIONS:
Overall Officials: Louise MONIOD, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Service de Gynécologie Obstétrique - CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No